CLINICAL TRIAL: NCT06148558
Title: A Twelve Week Clinical Study to Evaluate the Efficacy and Tolerability of a Sunscreen Moisturizer SPF 50+ in Women With Moderate to Severe Overall Photodamage
Brief Title: A Twelve Week Clinical Study to Evaluate the Efficacy and Tolerability of a Sunscreen Moisturizer SPF 50+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Revision Skincare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8674
Record Dates: First submitted 2023-11-14; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Anti-aging; Photoaging

STUDY DESIGN:
Intervention Model Description: Open label, 12-week study. 39 female subjects were recruited, 35 to 60 years, Fitzpatrick Skin Type I-VI, with moderate-severe overall facial photodamage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-Cell (Other)
  Interventions: Other: Sunscreen Moisturizer; Other: Gentle Cleansing Lotion; Other: Facial Moisturizer

INTERVENTIONS:
Other: Sunscreen Moisturizer — A provided anti-aging sunscreen moisturizer SPF 50 was used once a day.
Other: Gentle Cleansing Lotion — A provided Gentle Cleansing Lotion (Revision Skincare) was used 2x daily (AM/PM).
Other: Facial Moisturizer — A provided facial moisturizer (Goodier) was used 1x daily (PM).

SUMMARY:
The primary objective of this study is to evaluate the efficacy and tolerance of a moisturizer SPF 50+ when used over a 12-week time period by women with moderate to severe facial photodamage.

DETAILED DESCRIPTION:
This was a single center, single-cell, 12-week clinical trial on female subjects (Fitzpatrick Skin Type I-VI, evenly distributed) between 35-60 years of age with moderate to severe overall facial photodamage. All subjects were provided Revision Skincare Gentle Foaming Cleanser and Facial Moisturizer (Goodier Cosmetics) at the Screening visit after eligibility was confirmed. These products were used twice daily as instructed for a minimum 3 days prior to the Baseline visit (washout phase). At Baseline, subjects were given Sunscreen Moisturizer SPF 50+ to replace their Facial Moisturizer morning application. Subjects continued to use the Facial Moisturizer given at Screening in the evening.

Clinical grading assessments, full face images, Corneometer, Ultrasound, and subject self-assessment questionnaires were completed at each study visit (Baseline, Week 4, 8, and 12). Full face images were also completed post-application at Baseline.

A total of 34 subjects completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 35 and 60 years
* Women with Fitzpatrick skin type I-VI
* Subjects must have moderate to severe overall facial photodamage
* Subjects must have no known medical conditions that, in the investigator's opinion, may interfere with study participation.
* Subjects must be willing to provide verbal understanding and written informed consent.

Exclusion Criteria:

* Subjects who have demonstrated a previous hypersensitivity reaction to any of the ingredients in the study product(s).
* Subjects who are currently under a physician's care for a medical problem that, in the opinion of the Investigator or his designee, could affect the subject's treatment response.
* Subjects who are nursing, pregnant, or planning a pregnancy during this study
* Subjects who have a health condition and/or pre-existing or dormant dermatologic disease on the face
* Subjects who are not willing to avoid daily sun exposure on their face and the use of tanning beds or sunless tanning products during the duration of the study.
* Is currently taking or have taken within the listed time frame prior to the start of the study: Oral isotretinoin (Accutane®) within the last 6 months; Avita®, Differin®, Renova®, Retin-A®, Retin-A Micro®, Soriatane®, or Tazorac® within 3 months; Prescription-strength skin-lightening products within 4 months; Any anti-wrinkle, skin-lightening, or other product or topical or systemic medication known to affect skin aging or dyschromia within 2 weeks; Had a non-ablative laser (Including IPL) or non-ablative fractional laser resurfacing of the face and neck within 6 months
* Has any other condition that, in the opinion of the Investigator or his designee, could interfere with the subject's ability to use the treatment as instructed, alter treatment response, or affect their ability to complete the study.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Improvement in Clinical Efficacy Parameters at weeks 4, 8, and 12 versus Baseline | 12 weeks
  The primary efficacy endpoint will be Investigator Clinical Grading using a Modified Griffiths' 10-point scale. The scale ranges from 0 = none (best possible condition) to 9 = severe (worst possible condition). A decrease in score at post-baseline timepoints compared to baseline indicates an improvement. The parameters are fine lines (global face), wrinkles (global face), global hyperpigmentation (mottled and discrete), skin roughness (tactile), skin tone evenness (uniformity of skin color), overall photodamage, radiance (perceived glow), and skin firmness (tactile).

SECONDARY OUTCOMES:
Lack of significant increase in Objective Tolerability Parameters at weeks 4, 8, and 12 compared to Baseline | 12 weeks
  The primary tolerability endpoint will be the Investigator Tolerability Assessment of erythema, edema, and scaling/peeling of the face and neck. The 4-point scale ranges from 0 = none to 3 = severe. A decrease in score at post-baseline timepoints compared to baseline indicates an improvement.
Lack of significant increase in Subjective Tolerability Parameters at weeks 4, 8, and 12 compared to Baseline | 12 weeks
  The secondary tolerability endpoint will be the Subjective Tolerability Assessment of burning/stinging, itching, and tightness/dryness of the face and neck. The 4-point scale ranges from 0 = none to 3 = severe. A decrease in score at post-baseline timepoints compared to baseline indicates an improvement.

OTHER OUTCOMES:
Self-Assessment Questionnaire | 12 weeks
  The secondary efficacy endpoints will be the Self-Assessment Questionnaire on product efficacy and aesthetics. The 5-point scale ranges from 1 = completely disagree to 5 = completely agree. An increase in score at post-baseline timepoints compared to baseline indicates an improvement.
Improvement in skin density at weeks 4, 8, and 12 compared to Baseline | 12 weeks
  Ultrasound imaging of the left cheek will be used to measure skin density. An increase in value at post-baseline timepoints compared to baseline indicates an improvement.
Improvement in skin thickness at weeks 4, 8, and 12 compared to baseline. | 12 weeks
  Ultrasound imaging of the left cheek will be used to measure skin thickness. An increase in value at post-baseline timepoints compared to baseline indicates an improvement.
Improvement in skin hydration at weeks 4, 8, and 12 compared to Baseline | 12 weeks
  Corneometer measurements of the left cheek will be used to measure hydration content of the skin. An increase in value at post-baseline timepoints compared to baseline indicates an improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Skin Study Center, KGL LLC, Newtown Square, Pennsylvania, United States